CLINICAL TRIAL: NCT02507466
Title: Very Intensive Variable Repetitive AmbulatioN Training
Acronym: VIVRANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Thomas G Hornby, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00103739
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: locomotion
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 3 arm RCT - high intensity variable, high intensity forward, low intensity variable
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Variable high-intensity Training (Experimental): high intensity variable stepping exercise on a treadmill and overground
  Interventions: Behavioral: exercise
- Variable low-intensity training (Active Comparator): low intensity variable stepping exercise on a treadmill and overground
  Interventions: Behavioral: exercise
- Constant High Intensity Training (Active Comparator): high intensity constant (forward) stepping exercise on a treadmill and overground
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — Variable conditions of stepping practice

SUMMARY:
The overall objective of this subproject is to evaluate the individual and paired contributions of intensity and variability of stepping training on lower extremity (LE) function, health and community participation in patients with chronic hemiparesis post-stroke.

DETAILED DESCRIPTION:
The overall objective of this subproject is to evaluate the individual and paired contributions of intensity and variability of stepping training on lower extremity (LE) function, health and community participation in patients with chronic hemiparesis post-stroke. Using a RCT design/Intervention Efficacy paradigm, Aim 1 will investigate the independent and combined (paired) contributions of intensity and variability of stepping training on locomotor function, with secondary measures of health and community mobility. For Aim 2, we will evaluate the independent and combined effects of intensity and variability of stepping training on non-walking LE tasks. In Aim 3, we will evaluate the cost effectiveness of providing these interventions to accelerate motor recovery and health. Our central hypothesis is that results of this study will provide a theoretical foundation for implementation of physical therapy interventions which can facilitate short-term gains in locomotor function, and contribute to long-term improvements in health, function and participation through increased community mobility.

ELIGIBILITY:
Inclusion Criteria:

* history unilateral stroke > 6 months duration
* walks without physical assistance at speeds < 1.0 m/s

Exclusion Criteria:

* no other cardiopulmonary, metabolic, neurological orthopedic injury that may contribute to walking outcomes

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in peak walking speed | At baseline, following 8 weeks of training and a 2 month follow-up
  fastest comfortable walking speed overground

SECONDARY OUTCOMES:
Change in Functional Gait Assessment | At baseline, following 8 weeks of training and a 2 month follow-up
  dynamic balance activities
Change in 5X sit-to-stand transfer time | At baseline, following 8 weeks of training and a 2 month follow-up
  non-walking functional mobility task

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hornby, PT, PhD, Principal Investigator — RIC/NU
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300
- [Derived] Hornby TG, Henderson CE, Holleran CL, Lovell L, Roth EJ, Jang JH. Stepwise Regression and Latent Profile Analyses of Locomotor Outcomes Poststroke. Stroke. 2020 Oct;51(10):3074-3082. doi: 10.1161/STROKEAHA.120.031065. Epub 2020 Sep 4. PMID 32883192
- [Derived] Ardestani MM, Henderson CE, Mahtani G, Connolly M, Hornby TG. Locomotor Kinematics and Kinetics Following High-Intensity Stepping Training in Variable Contexts Poststroke. Neurorehabil Neural Repair. 2020 Jul;34(7):652-660. doi: 10.1177/1545968320929675. Epub 2020 Jun 6. PMID 32507027
- [Derived] Hornby TG, Henderson CE, Plawecki A, Lucas E, Lotter J, Holthus M, Brazg G, Fahey M, Woodward J, Ardestani M, Roth EJ. Contributions of Stepping Intensity and Variability to Mobility in Individuals Poststroke. Stroke. 2019 Sep;50(9):2492-2499. doi: 10.1161/STROKEAHA.119.026254. Epub 2019 Aug 22. PMID 31434543